# **Virginia Polytechnic Institute and State University**

# TOGETHER: A Couple's Model to Enhance Relationships and Economic Stability

**Unique Protocol ID: 15-960** 

**Study Protocol** 

**Date: March 29, 2018** 

A strong finances and families are the foundation of wellbeing for individuals, families, and communities. Low income families tend to experience chronic financial stress and are therefore, are at a higher risk for individual psychological and physical distress, relationship problems and dissolution, and parenting challenges, all of which in turn contributes to financial stress and economic instability. Financial stress and unstable economic conditions affect adults' individual well-being (e.g., substance abuse, depression and anxiety disorders), couple relationships (e.g., interpartner hostility, relationship dissatisfaction), and parenting, and children's emotional and physical health (Falconier, 2010; Kwon, Rueter, Lee, Koh, & Ok, 2003; Puff & Renk, 2014). Negative mental health outcomes can contribute to economic hardships through negative job outcomes. Recent research suggests that couple relationship education for disadvantaged couples could develop and sustain healthy relationships (Hawkins & Erickson, 2015). However, any efforts to intervene in the relationships and marriages of low income groups should directly address the chronic financial stress they experience and its permeating negative effects on different domains of their lives. Low-income couples might benefit more from a relationship education approach that helps them improve their relationship skills in the context of their financial stress and economically disadvantaged realities and connects them with the social services they need and with job/career enhancement resources that move their families towards economic stability and mobility. The interconnectedness of all of these factors influencing couple's relationships is important to address in a comprehensive intervention that integrates treatment components and takes into consideration the learning happening in other domains while focusing intervention in a specific treatment element or goal.

We target couples who live in Northern Virginia and Prince George's County and Montgomery County, MD. Even though these areas have high performing health and socio-economic outcomes for both the capital area and the nation, demographics have changed significantly in the past decade and disparities exist among subpopulations and low-income families. Overall high performing indicators may mask the true number of families that are seriously financially distressed and how racial/ethnic minorities are disproportionately more affected. This project is funded by the Department of Health and Human Services (HHS). Administration for Children and Families (ACF), Office of Family Assistance (OFA) under the Healthy Marriage and Responsible Fatherhood (HMRF) program. This project is developed and conducted by Project Director, Mariana Falconier, Ph.D. at Virginia Tech and Associate Director, Jinhee Kim, Ph.D. at University of Maryland. Both universities are collaborating for this project and University of Maryland is a subawardee of Virginia Tech. In addition, Virginia Tech has subcontracted with SkillSource Group, Inc. for delivery of the intervention and University of Maryalnd has contracted with Family Services, Inc. for delivery of Services. Services will be delivered at Virginia Tech, Family Service Inc. University of Maryland, and in agencies in which we have agreements to use their space (City of Bowie in Bowie, MD and Ebenezer Baptist Church, Alexandria, VA) The funding agency requires the grantee to have an independent local evaluator and for that purpose Virginia Tech has contracted with AVAR Consulting, which will be involved in the implementation and outcome evaluations. Avar Consulting as well as Dr. Falconier and Dr. Kim will only use the database without participants' identifying information to conduct their otucome evaluations The project employs a randomized control trial (RCT), in which 360 couples are assigned to the intervention group and 360 couples to a control group between June 1, 2016 and September 30, 2020. Our approach integrates three components (1) a 20-hour evidence-informed couple group program called TOGETHER workshop that integrates relationship education and financial literacy skills, (2) case management (assessment of participant needs, development of Individual and Couple Development Plan, referrals for social and mental health services, and referrals and coordination with job and career enhancement services. linking and coordination of all services as needed), and (3) job and career enhancement services for those who need the services. The main goals of this project are to promote healthy couple relationships and economic stability and mobility for low-income couples in Northern Virginia, Prince George's County, MD, and Montgomery County, MD. The main objectives are: 1) improve personal wellbeing; 2) improve

couple's relationship skills; 3) improve parenting and co-parenting; 4) improve financial literacy and capability; and 5) improve employability, job placement, and retention skills. Short-term outcomes of this project's core intervention are expected immediately after completion of the last session of the 20-hour relationship/financial education program (TOGETHER) whereas medium-term outcomes are anticipated six months after that last session. Expected measurable outcomes among program participants for objective 1 (improved personal well-being) include increased frequency of positive stress management, reduced psychological distress, decreased financial stress. Expected measurable outcomes for objective 2 (improved couple's relationship skills) include increased frequency of positive communication behaviors, increased frequency of positive conflict management behaviors, increased frequency of positive dyadic stress management, increased frequency of conjoint problem solving behaviors, increased satisfaction with couple's relationship, and increased comfort with financial styles and roles. Expected measureable outcomes for objective 3 (improved parenting and co-parenting) include increased frequency of positive parenting behaviors, increased closeness to children, and increased satisfaction with co-parenting. Expected measurable outcomes for objective 4 (improved financial literacy and capability) include increased financial literacy skills, increased financial self-efficacy, decreased use of alternative financial services, and increased financial management behaviors. Finally, expected measurable outcomes for objective 5 (improved employability, job placement, and retention) include decreased perceived barriers to employability, increased intentions and motivations for work, increased confidence in job skills, and increased employability, employment status, and retention.

The research team plans to use the study results to apply for future grants, write reports for the funding agency, submit manuscripts for publications, and disseminate results through conferences and public media appearances, as requested. Participants' identities will always be protected in any dissemination of study findings.

Target population in the proposed project is low-income couples, but any couple that wants to participate in the program will be accepted as long as they meet the eligibility criteria: residing in Northern Virginia and Prince George's County and Montgomery County in Maryland, married or cohabiting for at least a year, 18 years of age or older, and English-speaking. Exclusion criteria includes both partners being retired, physical domestic violence (defined as behaviors that frighten, terrorize, manipulate, hurt, humiliate, blame, often injure, and sometime kill, a current or former intimate partner) or feeling unsafe with partner in the last six months, current diagnosis of a severe psychiatric disorder that required hospitalization in the last 12 months, cognitive impairment, or/and severe untreated substance abuse disorder. Couples can participate as long as both partners consent to be part of the program.

To conduct the randomized control trial, 360 couples will be enrolled (180 from Northern Virginia and 180 from Montgomery County, Maryland) for the intervention group and 360 couples (180 from Northern Virginia and 180 from Montgomery County, Maryland) for the control group. Within each group (intervention and control), 20 couples will be enrolled in Year 1 (71/16-9/30/16), 100 in Year 2 (10/1/16-9/30/17), and 100 Year 3(10/1/17-9/30/18), 100 in Year 4 (10/1/18-9/30/19), and 40 in Year 5 (10/1/19-9/30/20).

Recruitment activities will be begin on June 1, 2016. Activities will include producing and distributing flyers, brochures, and posters and/or giving presentation in schools, churches, faith-based community centers, child support agencies, TANF offices, WIC agencies, Head Start programs, Healthy Start program, child welfare agencies, community centers, libraries, stores, barber shops, employment centers, Virginia Tech and University of Maryland clinics and cooperative extension centers, and community events. The Women's Center and Family Services Inc. will concentrate on marketing and recruitment efforts from the network of providers and partner organization they are part of. In addition, graduate students will be responsible for setting up social media outlets that will be used for marketing and recruitment purposes and posting calendars with program activities. The program will also be advertised through its own website (www.togetherprogram.org) and online ads.

The grant program manager will be responsible for overseeing all marketing and recruitment activities. These activities will be conducted by Virginia Tech and University of Maryland graduate student assistants and volunteers as well as designated administrative staff in The Women's Center and Family Services, Inc. (community partner agencies contracted for this project). The flyer and the brochure have been attached.

Low income families often experience greater social and economic challenges such as unemployment, poverty, low levels of education, poor job skills, and financial instability. They have limited access to resources to establish healthy relationships and economic stability due to limited social networks, skills and opportunities.

The target geographic areas in this proposal are Northern Virginia (VA) and Prince George's County Montgomery County, Maryland (MD), Even though these areas have high performing health and socio-economic outcomes for both the capital area and the nation, demographics have changed significantly in the past decade and disparities exist among subpopulations and lowincome families who struggle even more than before the last recession which occurred between December 2007 lasting until June 2009 (U.S. National Bureau of Economic Research). Although the median household income is high for Northern VA and Montgomery Co., MD (\$93,100 -\$122,238), the cost of living in these areas was 40% above the national average according to the 2010 U.S. Census and self-sufficiency standard for families has increased significantly in the last decades. For example, in Montgomery Co for a family of three the self-sufficiency standard doubled from \$32,016 in 1994 to \$68,086 in 2010 and contrasted markedly with the federal poverty level of \$17,600 for a family of three and the minimum wage job of \$12,792 for the annual full-time salary. Fairfax Community Action Board recommended using the number of people living in households with incomes below 200% as a better indicator of the level of need in those geographic areas as that indicator more closely approximates the level below which people have difficulty meeting their needs without some kind of assistance. In Fairfax Co 16.8% of residents and 18.3% of residents in Montgomery County live in households with earnings less than 200% of poverty, which indicates clearly the large number of families in this region that cannot meet their financial needs and that are at risk for individual, parenting, and relationship problems.

Couples interested in participating will be screened in person or over the phone by the trained project staff at the Northern Virginia Center of Virginia Tech, University of Maryland, Family Services, Inc., City of Bowie building or Ebenezer Baptist Church in Alexandria (VA), Staff must ask the couples for verbal permission before asking screening questions. If they meet eligibility criteria, they will be given an appointment with a case manager at any of the previously mentioned locations if the couple lives in Northern Virginia, Prince George's County or Montgomery County. MD. When the first appointment is made, participants will be provided with the information about program procedures. Potential participants will be offered the possibility of receiving a copy of the consent form by email or mail for their review prior to this appointment. This first appointment with the case manager is called "Intake and Enrollment Meeting." When the couple arrives for this meeting, the very first step that the case manager will take is describing the program TOGETHER in detail to the couple, providing them with an opportunity to ask any questions they may have. Once both partners in the couple say that they want to participate, the case manager will give each of them a hard copy of the consent form. The case manager will instruct each partner to read the consent form in detail and once again will invite partners to ask any questions they may have. The consent form will have every detail of the program including the risks and benefits. Additional simple instruction tools will be used to help participants understand the study procedures. Case managers will remind both members of the couple that their participation is voluntary and that at any time they may discontinue participation. Each partner will sign two copies of the consent, one for them to keep and another one for the program staff to store in a safe, locked cabinet.

The Program Manager of this project will be overseeing the process of obtaining and maintaining informed consents from subjects. The Program Manager will inform the Principal Investigator (Project Director: Dr. Falconier) and the Co-Investigator (Associate Project Director: Dr. Kim) of any problems that may arise. PI will also randomly check the process. In addition, an independent evaluator will be collecting data for evaluation of the program implementation and will alert the Principal Investigator and Co-Investigator of any deviations from the protocol for obtaining consent that is delineated in the Intake and Enrollment Protocol.

The consent process will take place in the offices of the Northern Virginia Center of Virginia Tech, the University of Maryalnd, Family Services, city of Bowie building, and Ebenezer Baptist Church in Alexandria, VA Inc. with the case manager that is meeting with the couple for the Intake and Enrollment Meeting. Family Services, Inc. Consent process will take place in private offices within each of those loactions with program case managers (all currently hired and supervised by Family SErvices, Inc.)

A case manager will hold an intake and enrollment meeting with every couple interested in participating in the program and that meets inclusion criteria. This meeting will take place before a couple participates in any activities of the TOGETHER program. During this meeting, the case managers will (a) explain the program procedures, obtain voluntary, informed written consent for program participation, (b) screen for domestic violence, (c) enroll participants and present overall program description, (d) collect and enter participant's demographic data in the online participant system for randomization, and (e) assign couples to the intervention or control group (see 5.1. for further details about this Intake and Enrollment Meeting).

When the project staff makes the first meeting appointments with case managers, the description of study procedures will be provided for potential participants to review the program prior to the first meeting. As noted earlier, potential participants will be given the opportunity of receiving by email or mail a copy of the consent form for them to review prior to the Intake and Enrollment Meeting (first meeting with the case manager). At the first meeting, the case manager will take the time to describe every aspect of the program and will give time for the couple to ask any questions they may have. Flowcharts and Schedules of Intervention and Control Group Couples will be provided to facilitate understanding of the program. Then the couple will be given time to read the consent form in detail and, again, ask any questions they may have. In the event that the couple says that they need more time to read the consent form, another appointment will be made to complete the intake and enrollment meeting. We will also be emailing an electronic copy of the consent form to those couples that want to receive such a copy before the Intake and Enrollment Meeting.

This study is being funded by a Healthy Marriage and Responsible Fatherhood (HMRF) grant by the Office of Family Assistance, Administration of Children and Families, U.S. Department of Health and Human Services. The funding agency requires all HMRF grantees to enter information into a secure system called the Information, Family Outcomes, Reporting, and Management system (nFORM). The information requested to enter is about (a) program operations (e.g., aggregated data without personally identifiable information on outreach and recruitment activities, enrollment numbers, staff qualifications and training, staff supervision and observation, and implementation challenges); (b) services (e.g., case management activities, workshop attendance, and referrals); (c) participants' contact information, demographics, and outcome measures. The funding agency also requires the use of tablets for collecting data from participants. This tablet will also be used to collect additional participants' outcome measures through Qualtrix. Please see Sections 5 and 8 for a further description of the nFORM system and data collection through Qualtrix.

See Intervention Group Flowchart for Participants document and Control Group Flowchart for Participants document in Attachments to follow each step of the procedure more easily. Besides nFORM and Qualtrix, two additional databases will be used to collect informaiton about participants and about program operations. One of them is called ICS database and is used to collect contact information about potential participants and screen them to see if they meet inclusion criteria before enrollment in the program. The section where identifying information such as participants' name, phone number or email address are stored separately from the answers to the screening questions. This ICS database is cleaned once a month so that all contace information is erased and only the number of participants that qualified or didn't qualify for the program can be counted. This ICS database complies with all VT requirements. It is an external service with prpoer SSL or similar encryption on the login and data collection pages. Only trained program staff (graduate assistants, programa managers, principal investigators, and quality assurance and operations coordinators will have access to this database. The second database is called Participant Trackign System (PTS). PTS is also compliant with all VT requireemnts for databases that collect participants' information as it is an external services with proper SSL or similar encryption on the login and data collection pages. PTS will be used for the purposes of automated randomization and scheduling meetings. The system is being developed and it may serve further functions in the future. We will request IRB permission first before it can serve other purposes. For the time being PTS will be used to collect contact information from participants to randomize according to place of residence and can help scheduling meetings. Trained program staff will have access to this database and this includes case managers, program manager, group facilitators, graudate assistants, quality assurance and program operations coordinators, and princiabl investigators. However, access will be restricted to each of these users so that participants' contact information is protected. PTS will be used for scheduling not only meetings for participants but also staff meetings (e.g., between case managers and group facilitators to discuss workhop concerns). PTS will not collect any information involved in the pre-,post- and follow up surveys (nFORM + Qualtrix) and therefore, it won't have the outcome data involved in data analysis. Same is true of the ICS database **Initial Contact and Screening** 

Individuals interested in participating in the program will dial a 1-800-number to the program staff or may visit the program at any of the program locations (Virginia Tech, University of Maryland, and Family Services, Inc.). Program staff will (a) collect contact information from the individual interested in participating, (b) describe the program and the potential compensation, (c) ask for verbal consent to proceed with screening questions, and (d) perform a 10-minute inclusion screening process of the potential participant and his/her partner. The program staff will speak with each partner during the call or visit if both partners are available. Otherwise, the program staff will collect information and screening information about both partners with the only partner that is present. However, when asking questions the staff will clarify that the caller is not required

to identify who of the two members in the couple does not meet elegibility criteria. Staff members administering the screening questions will obtain verbal consent to ask questions from the potential participant and will clarify that all screening data will be deleted after 30 days. All potential participants who are eligible after the initial screening and agree to participate will be scheduled for an Intake and Enrollment meeting with the case managers at Virginia Tech, The University of Maryland (UMD), Family Services Inc. (FSI), the city of Bowie, or Ebenezer Baptist Church in Alexandria, VA(see next section). The study procedure will be described and additional information will be sent upon request. Potential participants will be offered the consent form for them to review prior to the Intake and Enrollment meeting, given either in person or mailed to them upon request (Attachments: Initial Contact and Screening Script). ICS data will be saved in the ICS database.

Possibility of ICS Procedure online: Summary of Online Initial Contact and Screening (ICS) Procedure

Potential participants who are interested enrolling in the Together Program have the option of completing the screening with an ICS staff member online as well. If potential participants choose to complete the online screening, they can be directed to the screening in two ways: via a link an ICS staff member emails them after the potential participant and the ICS member review the Together Program Overview information together on the phone or via the Together Program website after the potential participant reviews the Together Program Overview information via the website.

Potential participants who obtain their information via the Together Program website will automatically be directed to the online screening page. Potential participants will review the Together Program Screening Information (please see below) prior to agreeing to the terms to continue with the online screening.

"Thank you for your interest in participating in TOGETHER program. You just read the overview of TOGETHER program, received an overview from one of our staff members over the phone, or watched our informational video.

Now you understand the program. We would like to ask you some questions about you and your partner to find out if our program can benefit you and your partner. Completing the questionnaire does not guarantee your eligibility. This screening process will take about 15 minutes to complete.

First, we will ask you to provide contact information and the best time to reach you and your partner in order to follow up. Then, we will ask some questions about you and your partner including your health and relationship. These questions address the issues of mental health, domestic violence, and substance abuse. Our program is not suited for everyone. These questions will help us to determine if you are eligible and if it is safe for you and your partner to participate in this program. It is important for you to have privacy when you are answering the screening questions. If you have any questions or would prefer to complete the screening process over the phone, you may contact the Together Program at 1-877-432-1669. You can choose to stop answering the questions if you do not want to participate.

Any identifiable information that you give us now will only be used to see if you are eligible to be in this program. After 30 days, we will destroy our records of your personal information. Should you have any questions about this study, or if you wish to complete the screening process via the phone you may contact the TOGETHER program at 1-877-432-1669.

By participating in this screening process, you are indicating that you are at least 18 years of age; the study has been explained to you; your questions have been fully answered; and, you freely and voluntarily choose to participate in the screening process."

Once potential participants have agreed to continue with the online screening, they will be prompted to enter information about themselves and their partner. This information includes their first and last names, phone numbers, and emails. Potential participants will also fill out their preferences for when they would like to be contacted, what location they would like to participate at, and the best days and times they are available for workshops. They are also asked to indicate how they heard about the Together Program.

Once potential participants fill out the demographic information, they will complete the online screening. Once they have completed the screening, they will receive the following message: "Thank you for completing the questionnaire! A trained staff member will review your answers and will be in touch with you by email or phone within 3 business days. We may contact you with additional questions. If you have any questions, you may contact the Together Program at 1-877-432-1669 or togetherscreening@gmail.com "

After potential participants complete an online screening, an email from "Together Screening" will be sent to the Together Screening Gmail Account with a notification message that a potential participant has submitted a survey. The notification will also give an overall score for the potential participant. The message will appear as the following:

"A potential participant has completed the online screening. This participant received a score of X Note: A score of 0 indicates there were no issues identified by the participant, any score 1 or above indicates participant has confirmed potential exclusionary criteria.

\*Please review response for completeness to ensure participant eligibility.

Please enter all information into ICS (using screening option 2) and contact the participant." Designated ICS staff (e.g., ICS Coordinator, Case Managers) will be responsible for checking the email account every 1-2 business days to review any recently submitted surveys.

Following this message will be a summary of all the potential participant's responses as well as the contact information they have provided. Designated ICS staff will be required to look through each of the responses to assess if there are any screening concerns that need to be addressed prior to calling the potential participant to schedule an Intake and Enrollment (IE) meeting. If there are no screening concerns, meaning that there is a score of "0," ICS staff insert the potential participant's contact and screening information into the ICS system and place the potential participant in the "Eligible and Further Action Needed" category. Once the potential participant is inserted into the ICS system, ICS staff will call to inform the potential participant that they are eligible for the program and to set up a day and time for the IE meeting.

If there are screening concerns, meaning that there is a score of "1" or higher, designated ICS staff will insert the potential participant's contact and screening information into the ICS system (refer to Appendix A for a list of questions taken directly from the online survey) but will need to follow up via phone call with the potential participant about the specific concerns. Designated ICS staff will refer to Section 9 in the Initial Contact and Screening Protocol for ineligibility requirements.

If a potential participant is ineligible due to their answers to the online survey (where no follow-up via phone call is needed), designated ICS staff will need to inform the potential participant that

they are ineligible for the program. Designated ICS staff will inform the potential participant via email and will provide the potential participant with referrals.

If ICS staff is unsure about specific concerns and/or questions, he or she should consult their supervisor.

Emails containing contact information and answers to screening questions will be deleted immediately after the information has been entered into the ICS database. The answers to screening questions collected through Qualtrix surveys will be deleted once a month. Intake and Enrollment Meeting, Part I

The first part of the Intake and Enrollment meeting will last 60 minutes. During the meeting, the case manager will (a) present a detailed program description and obtain voluntary, informed written consent for program participation from both partners; (b) conduct a formal assessment of domestic violence with each partner individually for 10 minutes (see Domestic Violence Protocol section and Domestic Violence Protocol in the Attachments); (c) enroll participants and collect contact information in nFORM; (d) assign couples to intervention or control group through an automated system of randomization that uses only state of residence (Maryland or Virginia) (PTS); (f) provide orientation about program procedures (one orientation for intervention couples and one orientation for control couples, participants will be given the "Welcome Letter and Instructions for Intervention Couples" or the "Welcome Letter and Instructions for Control Couples" and the "Control Group Flowchart for Participants" or "Intervention Group Flowchart for Participants"- See attachments); (g) describe participants with detailed explanation about payment procedures and VT and MD Tax requirements (providing VT and MD Tax requirements letters in attachmetns; and (h) direct and assist intervention and control couples to complete applicant characteristics survey nFORM and demographic information survey in a tablet (please see grant requirements regarding nFORM collection system)

#### Intake and Enrollment, Part II

The second part of the Intake and Enrollment meeting is different for intervention and control couples. For intervention couples (90 minutes; at VT, UMD, FSI, or by phone), the case manager will (a) provide an in-depth description of the study procedure (this will be supported by presenting couples with The Intervention Group Flowchart for Participants to enhance understanding - see this document in Attachments); (b) conduct a Needs Assessment in areas such as health care, employment, housing, childcare, education, legal barrier, income and financial, transportation, food, relationships, mental health, alcohol abuse, and substance abuse in order to determine which areas the couple needs support (see Needs Assessment document in Attachments); (c) schedule the individual and couple development plan (ICDP) meeting, progress meetings, and exit meeting as part of case management; (d) enroll couple in the eight-week TOGETHER workshop (20 hours; at VT, UMD, FSI or designated agencies/schools/churches) and a booster session which occurs three months after the completion of the TOGETHER workshop (3 hours: at VT or FSI); and (e) describe child care support and provide participants with the Child Care Support Letter (see attachments); and (e) explain the media release form and collect participants' signatures for those that agree to have their statements regarding the evaluation of the program be used in the media anonymously to advertise the program. The Schedule for Intervention Couples does not only indicate when and where the scheduled meetings and workshops take place, but also includes the incentives that couples may receive and the content of the meetings. All of these materials are included in the attachments. For intervention couples that do not wish to stay for the 90 minutes of the second part of the Intake and Enrollment meeting, the case manage will offer to conduct the Needs Assessment by phone with both partners at a later time that is agreed upon this meeting. At the end of the meeting the couples is compensated wtih \$40 (\$20/partner) in gift cards for participating in the Needs Assessment.

During part II for control couples, (90 minutes), the case manager will (a) provide a detailed description of the procedure for control group (this will be supported by presenting couples with The Control Group Flowchart for Participants to enhance understanding – see this document in Attachments); (b) oversee and assist couples complete pre-test surveys including the Pre-Program Survey (nFORM) and Pre-test Assessment (Qualtrics) (both surveys combined will take about 90 minutes - For content of assessments please see documents Pre-Program Survey nForm and Pre-Test Assessment in Attachments; (c) provide the couple their compensation in gift cards \$40 per couple (\$20/partner) for assessments; (d) ask partners to sign the Gift Card Receipt (see document in Attachments) after receiving the gift cards; and (e) schedule the couple for their post-test assessment meeting (in 8 weeks) and financial workshop/follow-up assessment (six months from the date of the post-test assessment meeting months). In the event that control couples cannot stay for this second part of the Intake and Enrollment meeting, they will be offered the possibility of completing the pre-program survey nForm and pre-test assessment in paper format or online. If the couple chooses to complete the survey and assessment in paper, they will be provided the questionnaires, the instructions to complete the questionnaire, and a selfaddressed envelope to mail the questionnaires. The instructions will explain that they will be mailed the gift cards once the guestionnaires are received and that they will be required to fill out a Gift Card Receipt (see document in Attachments). If the option is available and couples agree to it, they may receive the gift cards electronically once we have received the mailed questionnaires. If the couple chooses to complete the survey and pre-assessment online, we will be emailing to each partner the link and the individual passcode and we will be mailing the gift cards or provide them electronically, if this option is available and the couple agrees to it, once they complete the questionnaires.

#### **CONTROL COUPLES**

## **Control Couples: Post-Test Assessment Meeting**

Eight weeks after the Intake and Enrollment meeting, control couples will return to, VT, UMD, FSI or designated locations to meet with the case manager, and complete the Post Program Survey in nFORM and the Post-test Assessment in Qualtrics (both surveys combined will take about 90 minutes). ) The case manager will provide the couple their compensation in gift cards \$40 per couple (\$20/partner) for assessments and ask partners to sign the Gift Card Receipt Form (see document in Attachments) after receiving the gift cards.. Couples will be reminded about Financial Literacy Workshop (FLW) and follow-up assessment date. For couples that cannot attend the meeting in person, the questionnaires will be mailed to them with instructions on how to complete them and return them to the program in a self-addressed envelope included in the package (see Letter and Instructions for Post-Test Survey for Control Couples document and Post-Test Survey document (Post-Program Survey nFORM + Post-Test Assessment) in Attachment, Upon receipt of questionnaires by program staff, the gift cards and Gift Card Receipt Form will be mailed to the couple with instructions to complete the form and mail it back to the program staff in the selfaddressed envelope provided (see Letter and Instructions for Completion Gift Card Receipt Form in Attachments). If electronic gift cards are available and couples choose this option, the card will be emailed upon receipt of the questionnaires. Couples may also choose to complete the postsurvey and post-assessment online, in which case we will be emailing to each partner the link and their individual passcode and we will be mailing the gift cards or provide them electronically, if this option is available and the couple agrees to it, once they complete the questionnaires Control Couples: Follow-Up Survey/Financial Literacy Workshop

Six months after control couples will be invited to come 90 minutes before the Financial Literacy Workshop that will be offered for them. Trained program staff will provide tablets for these couples to complete the follow-up survey in Qualtrics before the beginning of the workshop. Completion of follow-up survey will take about 90 minutes. The trained program staff will provide the couple their compensation in gift cards \$80 per couple (\$40/partner) for assessments and will ask partners to sign the Gift Card Receipt Form. After the participants complete the follow-up survey, they will be invited to attend a three-hour Financial Literacy Workshop (FLW), led by

workshop facilitators at VT, UMD, FSI or designated locations. FLW is a three-hour financial management class to improve financial management knowledge and skills based on Money Smart curriculum by the Federal Deposit Insurance Corporation.

For couples that cannot attend the meeting in person, the questionnaires will be mailed to them with instructions on how to complete them and return them to the program in a self-addressed envelope included in the package (see Instructions for Mailed Follow-up Survey in Attachments). Upon receipt of questionnaires by program staff, the gift cards and Gift Card Receipt Form will be mailed to the couple with instructions to complete the form and mail it back to the program staff in the self-addressed envelope provided (see Letter and Instructions for Completion of Gift Card Receipt Form in Attachments). Couples may also choose to complete the follow-up survey online in which case we will be emailing to each partner the link and their individual passcode and we ill be mailing the gift cards or provide them electronically, if this option is avilable and the couple agrees to it, once they complete the questionnaires.

### **INTERVENTION COUPLES**

**Intervention Couples: ICDP meeting** 

Within two weeks of the Intake and Enrollment meeting, intervention couples will partake in an Individual and Couple Development Plan (ICDP) meeting with the assigned case manager at VT. FSI, UMD, or designated locations for 90 minutes. Based on the information collected in the Needs Assessment during the IE meeting, the case manager will create an Individual and Couple Development Plan with the couple that will include (a) setting individual and couple goals; (b) agreeing on action steps and establishing a realistic timeline to meet those goals; (c) discussing possible barriers participants might encounter; (d) providing referrals as part of the action steps to meet their goals (i.e., housing, TANF, health care, child welfare, child support services, mental health services, and job and career enhancement services). See the Individual and Couple Development Plan Form in Attachments. At the end of this meeting participants will be reminded of all of their scheduled appointments. If the ICDP includes a goal within the area of employment/career a first meeting will be scheduled for the partner in need of those services with an employment case manager to receive services at either the SkillSource Group, Inc. or a federally funded employment agency in Maryland depending on where the participant receives services in our program. In addition, the participant will be invited to sign a release to exchange information between the employment agency and our program so that information can be exchanged with the employment agency regarding information collected by our program (Couple's Needs Assessment and the Individual and Couple Development Plan) and the employment agency (employment/career services recommended and received, the participant's eligibility for those services, and the Employment Individual Plan). The signature of this release is necessary for the integration and coordination of services that are part of the present study. However, once the participant is referred to the employment agency, he/she becomes their participant and they are obliged to maintain confidentiality about their participants' information. The present study provides funding for (a) employment services for those participants that do not meet eligibility criteria to receive services funded through the Workforce Innovation and Opportunity Act (WIOA) or other state and local funding in those agencies and (b) for reporting all the employment/career services that participants referred from our program are recommended (Individual Employment Plan) and actually receive (Employment Services and Trainings Tracking Form) in such agencies. Since this study targets the low-income population, it is expected that most participants will meet eligibility criteria to receive services in those agencies funded through WIOA or state or local programs and not through this study. The Release to Exchange Information with Employment Agency is also necessary because the case manager will be sharing the needs' assessment and the ICDP and both documents relate to both partners and not just the one that may be receiving services at the employment agency. Therefore, both partners' consents are required to share those documents with the employment agency. Sharing these documents will allow the employment case manager to see what other referrals have been made for the couple. This is important information to avoid duplication of services as the employment agencies also have needs assessments and make referrals based on the individual's needs (see the Release to Exchange Information with Employment Agencies in Attachments, the Individual Employment Plan, Employment Services and Trainings Tracking Form, and the WIOA Eligibility Form). In

addition to paying for employment/ career services for participants that do not meet the eligibility criteria of for federally, state, or local funded employment programs, the current study provides fudning for two employment case managers, one for VA and one for MD. VA participants in need of employment services will be referred to an employment case manager working at SkillSource, Inc. MD participants in need of employment services will be referred to an employment case manager hired by UMD or FSI. that will assist participants in getting services (individual employment assessment and plan, trainings, and services) in WOIA employment agencies in Maryland. Employment case managers at VA and MD will be responsible for developing and/or collecting the individual employment assessment and plan and tracking all employment trainings and services that each participant receives). Even though it is desirable that both partners attend this ICDP meeting in person, the option will be giving to attend it by phone if partners can't attend in person. If partners choose to attend it by phone, the gift cards will be mailed to their home or emailed if this option is available.

**Intervention Couples: TOGETHER Workshop** 

Couples will begin the TOGETHER workshop at UMD, VT, FSI, or designated agencies, schools, or churches. TOGETHER is a 20-hour psychoeducational program for couples that supports the personal wellbeing, couple relationship, parenting, and financial literacy and management. TOGETHER was developed by Dr. Mariana Falconier (PI) and the late Dr. Hayhoe as part of the emerging interdisciplinary field that integrates relationship education with financial education (Falconier, 2015). TOGETHER adapted the Couples' Coping Enhancement Training (CCET) program developed by Dr. Guy Bodenmann (Bodenmann, 1997) and whose effectiveness in improving stress management, communication, and relationship satisfaction has been supported in various studies (Bodenmann & Shantinath, 2004; Lederman, Bodenmann, & Cina, 2007; Shaer, Bodenmann, & Klink, 2008) to financially distressed couples by applying CCET content to financial issues and incorporating financial education. The workshop aims at reducing financial stress and improving relationship functioning by providing couples with knowledge and skills on stress management, communication, conflict resolution and management, problem-solving, and financial management.

The TOGETHER workshop has 9 modules and is designed to be delivered in groups of four to eight couples for 20 hours: 8 weekly sessions of 2.5 hours each. Each session is co-led by two facilitators: a financial counselor and a couples therapist. Each session includes a warm-up activity, brief review of past session content and homework, presentation and practice of new content, summary of all contents covered in the session, and assignment of new homework. After each session, couples are assigned homework so that the skills learned in the session can be practiced between sessions. The TOGETHER curriculum has been pilot tested and results have been published in 2015 in the Journal of Marital and Family Therapy. FSI and TWC will hire couple therapists and financial counselors to provide these workshops. Couple therapists and financial counselors will be trained by Dr. Falconier and Dr. Kim.

The TOGETHER workshop will be offered at FSI, UMD, VT, or designated agencies, schools, or churches. There will be eight offerings in each facility per year. The workshop will be offered in eight sessions (2 hours and 30 minutes each) scheduled on the same day of the week and at the same time. Efforts will be made to offer the sessions in the evenings and on weekends to facilitate participation. Participants complete a 2 minute-session evaluation and a 2-minute homework evaluation within the time alloted to the session. In the last session they complete a 5 minute session evaluation+overall workshop evaluation within the session (see Session Evaluation questionnaire, homework evaluation questionnaire, and session evaluation and overall workshop evaluation questionnaire).

At the first TOGETHER session, couples will complete the Pre Program Survey (nFORM) and the Pre-test Assessment (Qualtrics) before the session begins. Completion of the Pre Program Survey and Pre-test Assessment will take about 90 minutes. For participants both surveys will be collectively referred to as "Pre-Test Survey". Partners will be instructed to complete these surveys in tablets provided by the group facilitators. Couples will receive compensations for

completing assessments in gift cards \$40 per couple (\$20/partner) and each partner will be required to sign and date the Gift Card Receipt Form upon receipt of the gift cards. TOGETHER session facilitators will oversee the completion of the Pre-Test Survey. Participants that fail to attend the first session of the TOGETHER workshop will be mailed the Pre-Test Survey for their completion (see in attachments these two documents: Instructions for Completion of Mailed Pre-Test Survey for Intervention Couples and the Pre-Test Survey (that shows the paper and pencil format for these two surveys combined: Pre-test Assessment and Pre-Program Survey). Participants will be instructed to return the completed surveys on the second session to receive their gift cards. Couples that wish to complete the pre-test survey online instead will be instructed on how to do so.

After the last (eighth) TOGETHER session, couples will start at either FSI, UMD, VT, or designated agencies to complete the Post Program Survey (nFORM) and the Post-test Assessment (Qualtrics). Surveys will take about 90 minutes. Participants will know these surveys as Post-Test Surveys and will complete them in the tables. Couples will receive compensations for completing assessments in gift cards \$40 per couple (\$20/partner) and each partner will be required to sign and date the Gift Card Receipt Form upon receipt of the gift cards. TOGETHER session facilitators will oversee the completion of the Post-Test survey. Participants that fail to attend the eight session of the TOGETHER workshop will be mailed the questionnaires with instructions on how to complete them and be given the gift cards (see in Attachments two documents: Instructions for Completion of Mailed Post-Test Survey for Intervention Couples in Attachments and the Post-Test Survey (that includes both surveys, the Post-Program Survey in nFORM and the Post-Assessment in Qualtrix). Couples that wish to complete the post-test survey online instead will be instructed on how to do so.

**Intervention Couples: Progress Meetings and Exit Meeting** 

Five weeks after the ICDP meeting, intervention couples will meet with the case manager for their first of five progress meetings (approximately five weeks between each progress meeting). The progress meetings occur at VT, UMD, FSI, or designated agencies. At each meeting, the case manager will (a) check progress towards goals established in the ICDP, (b) update the ICDP if necessary, (c) address barriers towards meeting ICDP goals, (d) check safety (e.g., presence of domestic violence), and (e) address any program issues (e.g., attendance to employment trainings, Two of these meetings will be in person and three over the phone and each of them will last around 30 minutes and will require the presence of both partners. However, the two in-person meetings will be conducted over the phone as well if the couple is unable to attend the meetings in person.

At the third progress meeting, case managers will provide the attendance incentives for the TOGETHER workshop. Case manager will provide couples with the gift cards \$80 per couple (\$40/partner) for perfect attendance (8 sessions), \$60 per couple (\$30/partner) for attending seven sessions, and \$30 per couple (\$15/partner) for attending six sessions. After providing the gift cards the case manager will ask both partners to sign and date the corresponding Gift Card Receipt form. If the couple does not attend the meeting in person. The gift cards will be mailed or provided electronically if this possibility is available and the couple agrees to it. Couples will have a final meeting with the case manager at VT, UMD, FSI, or designated locations 6 months after the last TOGETHER session, which will be approximately five weeks after the fifth case management progress meeting. At this exit meeting, the case manager (a) will make with the couple a final progress assessment toward the goals established by the ICDP, (b) will discuss with the couple their plan for continue working towards the ICDP goals, (c) will invite the couple to complete the follow-up survey in the tablets, (d) will provide \$80 in gift cards (\$40/partner) for completion of the follow-up survey, (e) will ask both partners to sign and date the Gift Card Receipt form, (f) will provide information about the TOGETHER program's Facebook group, and (g) will present the couple with a termination letter (see Termination Letter document in Attachments). If one or both partners cannot attend the meeting in person, the six-month followup survey will be mailed to them with instructions on how to complete them and return them to

the program in a self-addressed envelope included in the package (see Instructions for Mailed Follow-up Survey in Attachments). Upon receipt of questionnaires by program staff, the gift cards and Gift Card Receipt Form will be mailed to the couple with instructions to complete the form and mail it back to the program staff in the two self-addressed envelopes provided (see Letter and Instructions for Completion of Gift Card Receipt Form in Attachments). The couple will also be offered the possibility of completign this survey online for which instructions will be provided. If the couple chooses to complete this survey online, gift cards will be mailed or provided electronically if this option is available and the cople agrees to it.

Notes from all case management progress meetings and exit meeting with participants will be entered in the nFORM system. Data entered in these notes will not be used for data analysis by the investigators.

**Intervention Couples: Employment Services** 

At the ICDP meeting, case managers at VT, UMD, FSI, or designated agencies and will make referrals to Employment agencies for participants who need job and career enhancement services if needed after they review participants' work status, assess initial needs and job and education goals. Employment services will be provided by the SkillSource Group Inc, in Virginia and WIOA employment centers in Maryland. These agencies are the ones in Northern Virginia and Maryland that manage the federally funded WIOA that provides employment/career support services. The TOGETHER Project budget will be used to hire one employment case manager in each state (VA and MD) (two for the Project) and pay for the job assessment and trainings when participants are not qualified for the federal WOIA program (Workforce Innovation and Opportunity Act provides such services for eligible individuals for free) or other state and locally funded employment services. Case managers will contact employment case managers about the first appointment and communicate about the referral (clients) prior to the first meeting and as long as the Release to Exchange Information with the Employment Agency has been signed by both partners in the couple. Participants will be informed by the case manager and will receive reminders of the first appointment at SkillSource, Inc. and Maryland employment centers. In order to receive employment services and training, participants referred by the present study will have to become participants of those agencies. The release to exchange information signed by participants details the information that we will be exchanged between the two agencies (see earlier description). This exchange will allow for the integration of services as the employment case managers will review the couple's Needs Assessment and ICDP from case managers at the FSI and TWC and our program will have access to whether the participant is eligible for WIOA funded services (otherwise this study pays for services for non-eligible participants), the Individual Employment Plan, and the Employment Services and Trainings received. Qualified trainers will provide job development services, job related education and trainings in these agencies. However, neither the trainers nor the services are the responsibility of this study. We are only responsible for making the referral, collaborating in the exchange of necessary information for the coordination of services, and tracking the number and type of services recommended and received by participants. This integration and tracking of services will last for 6 months from the day of Post-Test Survey. After that day, participation in our study is concluded. However, participants can continue with the services with the employment agencies until their employment goals are met even though their participation in the TOGETHER program has concluded.

**Intervention Couples: Booster Session** 

completed by participants.

Intervention couples will be invited to a 3- hour booster session three months after completing the last session of TOGETHER workshop. These booster session will include up to 16 couples and will be co-led by a UMD or VT marriage and family therapy intern and a UMD or VT extension specialist. The booster sessions will occur at VT, UMD, FSI, or designated agencies and will offer an abbreviated version of the contents covered in the 20-hour TOGETHER workshop. Communication of Case Managers with Group Facilitators and Employment Case Managers

Employment case managers will not have access to the nFORM system or any of the surveys

Communication among case managers and employment case managers will only take place if there is a release to exchange information signed by each member of the couple. Providers will communicate primarily through conference calls or in-person meetings. There will be weekly conference calls, or, if possible, in-person meetings (1) between case managers and group facilitators, and (2) between case managers and employment case managers. During these meetings, attendees will go over the list of project participants that they share and will update each other about relevant issues that need to be taken into consideration when working with these couples/individuals. Should communication be necessary beyond the scheduled meetings with the case manager, any of the employment case managers or group facilitators can email and/or make a phone call to the case manager if there is an issue related to the participants that cannot wait to be addressed in the following scheduled meeting. Similarly, the case manager will be able to contact the group facilitators and/or employment case managers if needed before the next scheduled meeting. In all of these communications, only participants' ID (nFORM ID) will be used in any records. Case manager communication with group facilitators and employment case managers have to be entered in the nFORM system that tracks all case management operations. **Domestic Violence and Child Maltreatment** 

All the program staff that interacts with program participants will be receive a three-hour training to learn to identify, assess, and response to situations of domestic violence. In addition, the funding agency requires the program staff to report to the corresponding local authorities any situation of maltreatment. Therefore, the training for program staff will also include information on what constitutes child maltreatment and when and how to report any suspicion of child maltreatment.

Regarding domestic violence, a pre-screening for domestic violence will take place in the Initial Contact and Screening stage before participants are enrolled in the program. Then, later, after enrollment but before randomization and entering participants' information into the nFORM a structured screening for domestic violence will take place so that cases of domestic violence can be referred to appropriate services and participation in the program is discontinued. This structured screening involves an individual 10-minute meeting with each partner, during which each will be asked questions about any incidents of physical, sexual and/or psychological violence that have occurred in their relationship. Each partner will also be asked about whether or not they feel threatened by their partner, and whether or not they feel safe in participating in the program with their partner. Additionally, each partner will be asked about his/her willingness to commit to safety and no violence, and his/her willingness to learn strategies to de-escalate conflict between them in a safe way. Based on the participants' responses, a determination will be made regarding the couples' participation in the program. If both partners provide responses that indicate a lower risk for domestic violence, then the decision will be made that they can continue participating in the program with no referral for additional services to directly address domestic violence. However, if either partner provides:

- 1. Responses indicate the presence of domestic violence in the current relationship
- 2. Responses describe minor domestic violence, including pushing, shoving
- 3. Responses describe infrequent domestic violence, and/or incidents which occurred more than one year ago
- 4. Responses indicate no weapons in the home

The decision will be made that the couple may participate in the program, and they would be referred to services that directly address domestic violence. This decision will be made if both partners also indicate a commitment to no violence and both feel safe participating in the program with each other. In these instances, partners would have to provide permission for the case manager to consult and coordinate with the domestic violence provider, to determine treatment progress and to verify treatment completion. The permission will be provided by signing a release to exchange information with domestic violence services (see Release to Exchange Information with Domestic Violence Agency in Attachments). If further or worsening violence occurs with the first eight weeks of the program, the couple would be asked to discontinue participation from the program (see Termination Letter Due to Safety Issues).

Request to discontinue participation in the program and referral to domestic violence services may also occur at any point in the participation in the TOGETHER program beyond the initial

structured screening at the Intake and Enrollment meeting. This would be situations when the case manager has found that it is unsafe for one or both partners to continue participation in the program. Case manager may find out about the presence of domestic violence by him/herself or through the suspicions of other program staff that request the case manager to assess for the presence of domestic violence. If during the course of screening for domestic violence, an immediate emergency or concern for the safety of either partner or staff occurs, case managers will be instructed to contact police.

The consultant expert on domestic violence, Dr. Norman Epstein, has provided and will continue providing his expert opinion regarding the Domestic Violence and Child Maltreatment protocol, staff training, and issues that may arise during program delivery (see Domestic Violence Protocol and the Child Maltreatment Protocol in Attachments).

For the purposes of making prompt referrals, VT has signed MOUs with FSI, TWC, and the Fairfax County Office for Women and Domestic and Sexual Abuse Services.

Program Termination

Individuals may terminate their participation in the program for several reasons. They may have participated in the exit meeting concluding their participation in the TOGETHER program. In such instances, a termination letter will be mailed (see Termination Letter in Attachments). Individuals may discontinue participation and failed to respond to case manager's contact attempts. In those situations, participatns may be invited to withdraw if they are no longer interested in participating in the TOGETHER program. In that case a letter will be mailed to participants (see the following three documents in Attahcments: the Letter for Potential Termination of Program Participation for Mailed Follow-up Surveys Not Returned, the Letter for Potential Termination of Program Participation for Intervention Couples when Missed Appointments, and the Participant's Program Withdrawal Letter in Attachments). The case manager will also complete a Case Management and Employment Services Summary form for every couple. This form does not contain participants' identifying information but only participants' ID. The form will be entered by graduate assistants in VT or UMD into the database to be submitted to AVAR for data analysis.

Individuals may also be requested to discontinue participation in the program if it is no longer safe for one or both partners to continue participating in the TOGETHER program (see Termination Letter due to Safety Issues in Attachments).

We are describing in detail all the data that will be obtained from participants. However, only the non-identifiable data will be used for data analysis of program outcomes by AVAR (the local evaluator) and Dr. Falconier and Dr. Kim (PI and Co-PI). The non-identifiable database will be made up of all surveys completed by the participants (Applicant's Characteristics, Demographic Information, Pre-Test Survey, Post-Test Survey, Follow-up Survey, TOGETHER Homework Evaluation, the Evaluation of the TOGETHER session) and the Case Management and Employment Services Summary data completed by the case manager. The rest of data collected from participants will not be part of the database for analysis or used for data analysis. These data are only collected with the purpose of providing services to participants.

The funder (ACF) requires the program performance evaluation data collection using nFORM. We are required to enter the information about (1) program operations (e.g., outreach and recruitment activities, enrollment, staff qualifications and training, staff supervision and observations, and implementation challenges), (2) services (e.g., case management activities, workshop attendance, and referrals) in nFORM. Service information will be entered within hours no later than 24 hours after session. If any notes or log have been written down, the paper will be shredded or kept in a locked cabinet after the data is entered. Additionally, we will use paper files to collect program operation and services data and keep in the locked cabinet.

Program operations will be used as aggregate forms and no personally identifiable information will be included. These data will be used to generate required grant reports and to improve the implementation of the project. However, any personally identifiable information will never be linked to participants' surveys for the purpose of research.

Besides nFORM and Qualtrix, two additional databases will be used to collect informaiton about participants and about program operations. One of them is called ICS database and is used to collect contact information about potential participants and screen them to see if they meet inclusion criteria before enrollment in the program. The section where identifying information such as participants' name, phone number or email address are stored separately from the answers to the screening questions. This ICS database is cleaned once a month so that all contace information is erased and only the number of participants that qualified or didn't qualify for the program can be counted. This ICS database complies with all VT requirements. It is an external service with prpoer SSL or similar encryption on the login and data collection pages. Only trained program staff (graduate assistants, programa managers, principal investigators, and quality assurance and operations coordinators will have access to this database. The second database is called Participant Trackign System (PTS). PTS is also compliant with all VT requireemnts for databases that collect participants' information as it is an external services with proper SSL or similar encryption on the login and data collection pages. PTS will be used for the purposes of automated randomization and scheduling meetings. The system is being developed and it may serve further functions in the future. We will request IRB permission first before it can serve other purposes. For the time being PTS will be used to collect contact information from participants to randomize according to place of residence and can help scheduling meetings. Trained program staff will have access to this database and this includes case managers, program manager, group facilitators, graudate assistants, quality assurance and program operations coordinators, and princiapl investigators. However, access will be restricted to each of these users so that participants' contact information is protected. PTS will be used for scheduling not only meetings for participants but also staff meetings (e.g., between case managers and group facilitators to discuss workhop concerns). PTS will not collect any information involved in the pre-,post- and follow up surveys (nFORM + Qualtrix) and therefore, it won't have the outcome data involved in data analysis. Same is true of the ICS database

As noted in the procedures section for online ICS, the screening information collected through Qualtrix will be erased once a month.

**Case Intake Information** 

PTS: After the consent form is singed by participants, the case manager will open a new participant file in PTS and will enter all of the participants' contact information to be able to randomize participants in the automated system and to schedule meetings with case managers in the PTS system.

nFORM: After the consent form is signed by participant and randomization takes place, the case manager will open up a new participant file in the nFORM system and enter all of the participants' contact information, including if they are an intervention or a control group couple. This new client information will be used only for program management, and is not linked to any of the couples' other survey data. Additionally, nFORM personal information data cannot be downloaded.

Paper: The case manager will also create a hard case file for each couple at the first intake and enrollment meeting. He/she will put the couple's consent form in the file, and label it with their ID number on the tab. The case files will be kept in a locked drawer in a locked office in either the WC or FSI. When a case is no longer active the case manager will take the papers out of the file in the same order, and scan the files. These scanned files will be saved under the couple's ID numbers. They will then be stored on a secured university hard drive. The hard copies will be shredded. Case Management Information

PTS: case management meetings will be scheduled in PTS

nFORM: All case management contacts and referrals will be recorded in the service entry of nFORM under the client ID. Service entry forms contain with information about date, case manager's name, types of meeting, the length of visit, and service notes

Paper: Intervention Group Participants will receive case management including Needs Assessment, Individual and Couple Development Plan (ICDP), five progress and one exit meetings. Needs Assessment and ICDP forms will be created by the case manager. These forms will be stored in the couple's case files; a copy will be provided to the couple, too. These forms will contain only couples' ID numbers but not any personal or identifying information. TOGETHER Workshop

TOGETHER workshop facilitators will take notes about their own observations of couples' needs, concerns, special circumstances, and progress toward goals after each session every week. This note contains only client ID but no identifying information.

Also facilitators will collect the session evaluation questionnaire to improve the workshop implementation. The session evaluation questionnaire does not contain any identifying information or client ID.

**Employment Services (see also 5.1.)** 

Employment Case Managers hired by FSI, or SkillSource Group, Inc. will develop an Individual Employment Plan and will provide job and career enhancement services for participants who are interested in receiving such services. The Release to Exchange Information with Employment Agencies will allow our program staff to have access to the Individual Employment Plan as well as the employment services and trainings that each participant referred from our program has completed.

Process evaluation information regarding the numbers of referrals, intake, Individual Employment Plan Development, job assessments completions, job education and training attendance and

completions, and other job related services rendered will be tracked. Employment case managers will share these information but they will contain only ID number but no personally identifying information.

**Exchange of Information Among Providers (see also 5.1.)** 

During the course of the TOGETHER program the case manager may need to communicate with the employment case managers (SkillSource Group and MD employment centers) and/or providers of services (e.g., domestic violence agency) that the couple has been referred to outside the TOGETHER program. In both situations, the case manager will have to obtain releases from both members of the couple even if the services are just for one member of the couple. Authorization to release information is needed from both partners in the couple as most of the meetings and notes by the case manager involve and are about both partners in the couple. The purpose of obtaining a release form is for coordination of services with the other provider. It is an exchange of information, allowing communication to flow between the indicated parties in both directions. However, the case manager should not disclose any confidential information about the couple beyond what is strictly necessary to coordinate services. Releases may be rescinded by the client at any time.

**Case Management Data for Analysis** 

Once a couple's file is terminated the assigned case manager will complete a Case Management and Employment Services Summary form (see this document in Attachments). This form will include: the number of case management meetings attended, the types of referrals for the couple and family members, and the employment services recommended and received by each partner if there was a need for employment services. Data from this form will be entered by VT or UMD graduate assistants in the database that AVAR will receive with the data from participants. This database will be used for data analysis by AVAR and program investigators and does not contain any identifying information.

**Independent Evaluator Process Evaluation** 

AVAR consulting will review documents such as work plan, protocols, surveys, conduct key personnel interviews, on-site observations, conduct focus groups with participants, and access the Qualtrics and nFORM downloaded non-identifiable data and the non-identifiable case management and employment services summary data.

**Focus Group by Independent Evaluator** 

An experienced researcher will conduct focus groups of program participants about their experiences and satisfaction with the TOGETHER program. Intervention couples, specifically, will also be asked within these focus groups about their experience with the integration of program services. The focus group will be conducted once annually at each intervention sight, and will include 8 individuals (4 couples). The inclusion criteria for the group is that the individual has enrolled in the TOGETHER project and was assigned to the intervention group, completed at least one assessment, and attended at least four TOGETHER sessions. An experienced note taker who will accompany the focus group facilitator will transcribe the discussions within each focus group. Focus groups will last 60 minutes. Participant selection for the focus groups will not be known at the time of enrollment, but it will be indicated to the participants that they might be selected for the focus group and notified of their participation within three weeks of participation. Risks are minimal in that no sensitive or personal information will be requested. However, participants will be asked about their experience in the project. The group might experience some discomfort in re-living an emotional experience. The focus groups will be held at the program sites; therefore, there will be resource persons available to assist in these instances. The benefits of participation in the focus groups are not for the individual participants, but will benefit the overall target population in that their feedback and suggestions will be used to improve project processes and implementation. At the time of the focus groups, during the opening, participants will be reminded that there participation is voluntary, that they can refuse to answer any question, and may withdraw from participating at any time without losing any services or rights to participation in other aspects of TOGETHER or at the program site. The focus group facilitator

will ask the participants for verbal consent to proceed with the group before beginning the formal discussion of topics/questions.

Notes from the focus group will be word-processed and analyzed by trained raters and coders. From the time the focus group transcriptions are created until three years beyond the end of the grant, all electronic versions of the notes will be filed in the evaluator's password-protected electronic files and all hard copies of notes will be maintained in locked file cabinets at the evaluators' site. At the end of the three-year time-period post-grant, the electronic files will be permanently deleted from computers, servers, or the cloud, and printed copies of the notes will be shredded.

There might be an emotional risk to participants. Although the instruments, session activities, homework assignements, and material presented at the TOGETHER program that will be used in this study have been widely used in research and intervention and psychoeducational programs without concerns, some participants might experience feelings of discomfort (e.g., sadness or anger) as a result of completing the questionnaires, participating in the session activitivies, completing homework assignmens, and learning about the content presented at the TOGETHER program. To address any emotional of these emotional issues that may arise, case managers will make appropriate referrals for therapy or added required services. For domestic violence issues, see 5.2.

Anticipated benefits to study participants include increased frequency of positive stress management, reduced psychological distress, decreased financial stress, increased frequency of positive communication behaviors, increased frequency of positive conflict management behaviors, increased frequency of positive dyadic stress management, increased frequency of conjoining problem solving behaviors, increased satisfaction with couple's relationship, increased comfort with financial styles and roles, increased frequency of positive parenting behaviors, increased closeness to children, increased satisfaction with co-parenting, increased financial literacy skills, increased positive attitude toward financial management, increased financial management behaviors, decreased perceived barriers to employment, increased intentions and motivation for work, increased confidence in job skills and increased employability, employment status and employment retention. In addition, participants will receive incentives in the form of gift cards for their time in the program, referrals to community resources, and job and career services (e.g., job education and trainings).

The funding agency, Administration for Children and Families (ACF) will collect the data utilizing a management information system, called nFORM. nFORM is web-based and does not require users to download any applications or program any code. As ACF's contractor, Mathematica will analyze the administrative performance measures data collected by the all grantees, including the current project. Mathematica has received a waiver of consent from the New England Institutional Review Board to analyze these data without specific consent from grantee clients to do so. Standardized performance measurement and reporting across HMRF grantees will enable ACF to track programming outputs and outcomes across programs to inform HMRF program design, operation, and oversight.

The project's independent evaluator, AVAR consulting, will have access to the data (downloaded from nFORM and Qualtrics) for research data analysis without any identifying information.

Through the data entered in the nFORM system the Office of Family Assistance (Administration of Children and Families, US Department of Health and Human Services will have access to identifiable data. However there are two separate systems in nFORM, one that collects identifable information for case management and service delivery and one for non-identifiable outcome data about participants (Applicant's Characteristics, Pre-Test Program Survey, Post-Test Program Survey).

After the participants have completed the consent form, enrolled in the program, and assigned on intervention or control groups randomly, case managers will generate the client ID by filling out the intake form in the nFORM. These nFORM IDs instead of identifying information will be used for all assessment surveys completed by participants and any other data for program operation and services.

Case managers will collect and access personally identifiable information (PII) such as nFORM client information, consent forms, receipts, and release forms. These data include clients' identifying information such as name, phone number, email address, and home address and aspects about clients' involvement in the program for service delivery and program operation. nFORM Client information containing PII will not be downloadable or exportable. Data containing PII in a paper form will be separate from participants' all other documents such as needs assessment, Individual and Couple Development Plan, and case meeting notes which will contain only client ID. However, case managers will not have any access to the survey assessments data that will be used for analysis.

Two additional databases will be used. One for potential participants that are screened (to see if they meet inclusion criteria) over the phone or in person before enrollment in the program. This is called the ICS database. The section where identifying information such as participants' name, phone number or email address are stored separately from the answers to the screening questions. This ICS database is cleaned once a month so that all contace information is erased and only the number of participants that qualified or didn't qualify for the program can be counted. This ICS database complies with all VT requirements. It is an external service with prpoer SSL or similar encryption on the login and data collection pages. Only trained progra staff (graduate assistants, programa managers, principal investigators, and quality assurance and operations coordinators will have access to this database. The second database is called Participant Trackign System (PTS). PTS is also compliant with all VT requireemnts for databases that collect participants' information as it is an external services with proper SSL or similar encryption on the login and data collection pages. PTS will be used for the purposes of automated randomization and scheduling meetings. The system is being developed and it may serve further functions in the future. We will request IRB permission first before it can serve other purposes. For the time being PTS will be used to collect contact information from participants to randomize according to place of residence and can help scheduling meetings. Trained program staff will have access to this database and this includes case managers, program manager, group facilitators, graudate assistants, quality assurance and program operations coordinators, and princiapl investigators. However, access will be restricted to each of these users so that participants' contact information is protected. PTS will be used for scheduling not only meetings for participants but also staff meetings (e.g., between case managers and group facilitators to discuss workhop concerns). PTS will not collect any information involved in the pre-,post- and follow up surveys (nFORM + Qualtrix) and therefore, it won't have the outcome data involved in data analysis. Same is true of the ICS database

Program staff at Virginia Tech and University of Maryland will keep paper data containing PII such as the list of gift cards recipients and child care vouchers (see section 9.1) separate from any program evaluation data in the locked cabinet.

However, only PI, Associate Director, and Program Manager will have an access to both the survey data with client IDs and identifying information that can be linked to the IDs.

nFORM is hosted and maintained by Mathematica and all data are stored on secure servers behind Mathematica's firewalls. Safequards used to protect sensitive data stored within the nFORM system are consistent with the Privacy Act, the Health Insurance Portability and Accountability Act, the Federal Information Security Management Act, and National Institute of Standards and Technology security and privacy standards. Identifiable data will be encrypted at all times (in transit and at rest) using cryptographic modules that are compliant with Federal Information Processing Standard 140-2, and will be securely deleted from the system when no longer needed. Access to the nFORM system will be controlled via multifactor authentication mechanisms and will be limited for both grantee and Mathematica staff. In addition to these nFORM-specific procedures, Mathematica has extensive corporate administrative and security systems to prevent the unauthorized release of personal records, including state-of-the-art hardware and software for encryption that meets federal standards, other methods of data protection (e.g., requirements for regular password updating), and physical security that includes limited key card access and locked data storage areas. Mathematica also requires every employee to sign a pledge to protect the privacy of data and client identity, and breaking that pledge is grounds for immediate dismissal and possible legal action.

All program staff will be trained in protection of sensitive and/or confidential information as part of their training on data collection. Examples of data that will be collected include downloaded online survey data and interview responses. Those data containing identifying information will be separate from participant' case files, which include participants' needs assessment, individual and couple development plan meeting (IDCP), and case management notes. The case files are for active cases and are only identified by client case number. The files will be filed in folders with dividers in locked cabinets at VT, UMD, or FSI. There will be one file per couple. The couple's ID number (no identifying information) will be printed on the tab of each file folder. The following information will be kept in each case file, each identified only with the client ID number to help protect clients' identifying data. The case files will have each couple's ID number written on the tab (no identifying information will be included in or on the case file). The files will be stored in locked file cabinets at VT, UMD, or FSI.

Downloaded nFORM and Qualtrics data will be stored in the password protected computers at Virginia Tech and University of Maryland. All other data collected in papers will be stored in a safe, locked cabinet at Virginia Tech. Access to electronic data will be limited and based on staff responsibilities and will be securely protected.

The project includes a program performance evaluation plan for the collection, management, and analysis of nForms data about participants and program operations and a funded activities evaluation plan developed in collaboration with an independent local evaluator (AVAR, Consulting). The funding agency, ACF expects grantees to conduct grantee-specific evaluations, called "local evaluations" to answer one or more grantee-specific research questions. The purpose of these evaluations is to learn from programs in order to improve future programming. Local evaluations must be designed to help inform future programming and expand the evidence base. Local evaluations must be conducted by an independent evaluator, referred to as the "local evaluator." The funding agency requires local evaluator with experience in conducting rigorous evaluations. Avar Consulting, Inc., an independent policy research firm specializing in attitude-behavior research, program evaluation, and survey methodology signed a letter of commitment to conduct our local impact evaluation.

AVAR consulting will conduct key personnel interviews, on-site observation, focus groups with participants, and access the data exported from nFORM and Qualtrics (without identifying information). All the evaluation related data will be also stored on the AVAR consulting, independent evaluator's secure server and handled in accordance with the NIST SP800-53 security procedures.¬¬ AVAR consulting will conduct focus group to collect qualitative data about participants' experiences and satisfaction with the TOGETHER program. The local evaluator's IT facilities and data security procedures have been rigorously inspected and approved by the

Centers for Medicare and Medicaid (CMS) for handling sensitive data with individual personal identifiable information (PII). Having conducted numerous surveys for various federal agencies, the local evaluator has also established rigorous procedures to ensure data confidentiality, such as separating PII data from survey data; transferring PII data only through password protected FTP (File Transfer Protocol) sites, CDs, or USB drives; and forbidding staff from saving PII data on individual desktops or laptops. All the relevant evaluator staff have received data confidentiality training and signed a confidentiality pledge.

AVAR consulting staff and Dr. Falconier (PI) and Dr. Kim (Co-PI) as well as other UMD and VT program staff involved in data analysis.

Data collected in paper format wil have been completely entered by the time participants' participation is terminated. Electronic identifiable data will be password protected and kept in VT secure hard drive and it will be deleted two years after funding for this study has been concluded (at present the expectation is to be funded by ACF until 9/30/20. All electronic non-identifiable data will be kept for 15 years for data analysis.

Intervention and control couples will be paid \$160 for completion of assessments (Pretest: \$40 (\$20/partner), Post-test: \$40 (\$20/partner), Follow-up: \$80 (\$40/partner)). Additionally, intervention couples will be given \$40 gift certificate (\$20/partner) for a local grocery store for attending the Needs Assessment meeting with the case manager. Lastly, after completion of the TOGETHER workshop, intervention couples will receive an incentive, \$30-\$80 in gift cards.

To help remove barriers to participation in the program of intervention couples, childcare support (\$280/couple) are budgeted to recruit and engage participants with children ages below 12, unless the program is able to provide child care onsite during the workshop. Program staff will provide Childcare Reimbursement forms to participants to be redeemed. At a later date a check will be sent directly to the person(s) providing the childcare while the participants attend program sessions and meetings. The total amount for childcare will not exceed \$280 per couple, and are viewed as a cash equivalent and are therefore taxable. Therefore, In order to obtain childcare reimbursement, participants must complete both the W-9 for tax reporting and the Child Reimbursement forms, and obtain the signature of the childcare provider. They must then submit these completed forms to their case managers. The child care provider must be a licensed child care provider.

Caseworkers will determine participant eligibility to receive childcare support at progress and exit meetings. If eligible and if no child care is provided for free by the program onsite during the workshops, caseworkers will issue the Childcare Reimbursement form and a W-9 form to the participants. Participants will secure childcare while they are attending eligible training/educational events or meetings as a direct result of participating in the TOGETHER project. A new W-9 form must be completed and submitted to the caseworker for each new provider; if a provider provides services on more than one occasion, he/she need only submit the W-9 form once. The caseworker will verify the validity of reimbursement request, record receipt of the reimbursement and W-9 forms in the Couples' Childcare Log, and send the completed forms to Dr. Mariana Flconier at Virginia Tech and Dr. Jinhee Kim at University of Maryland (Maryland participants), the Principle investigator of this project, at Virginia Tech. Once received, the forms will be recorded on the "TOGETER-Childcare Request and Reimbursement Lob." Information stored on the log includes: date request received, the ID number of the participant(s) to which the reimbursement form was issued, the name and address of the childcare provider, and the amount of reimbursement requested. The program manager will first verify that the \$100 limit has not been reached for that participant, and then mail the check to the childcare provider directly to the address provided on the W-9 form. Upon receipt, childcare providers are requested to complete, sign, and return the reimbursement receipt form in the stamped return envelope (both supplied with the check).

Only the incentive for the completion of TOGETHER workshop will be prorated. Depending on the number of Workshop sessions that both partners attended:

8 sessions: \$80 gift card (\$40/each partner) 7 sessions: \$60 gift card (\$30/ each partner) 6 sessions: \$30 gift card (\$15/each partner)

Participants receive compensation only for completion of assessments if they actually complete them, for attendance to ICDP meetign if they attend it in person or by phone, and for TOGETHER workshop attendance if they actually both partners attend the specified number of sessions.